CLINICAL TRIAL: NCT01963585
Title: Evaluating the Capacity of High-sensitivity Serum CRP Levels to Predict Bronchial Hyper Responsiveness in School Age Children
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0200-11
Record Dates: First submitted 2013-10-13; First posted 2013-10-16 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Hyperreactive Airway
Keywords: C reactive protein; Airway hyperreactivity; Body mass index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Negative metacholine: Healthy control
- Positive metacholine: Hyperreactive airway disease - study group

SUMMARY:
Background:

Bronchial hyper responsiveness (BHR) assessed by methacholine challenge test (MCT) may aid in the diagnosis of asthma, while negative MCT can help to exclude the diagnosis. Laboratory measures that predict the results of MCT are expected to reduce the number of procedures. The possible capacity of High sensitive C-reactive protein (hs-CRP), a marker of systemic inflammation, to predict negative or positive MCT in children has not been evaluated.

Aim: to evaluate the capacity of hs-CRP to predict positive or negative MCT in school aged children and to compare it with markers of airway inflammation: Fractional exhaled Nitric Oxide (FeNO) and markers of allergic sensitization (IgE and peripheral blood eosinophils).

Design: Prospective study evaluating these parameters in patients with positive and negative MCT.

Participant selection: The study population included subjects (age range 6 to 18 years) referred for Methacholine Challenge Test (MCT)

Sample size: 130 participants in the two groups. Intervention: Each subject will undergo evaluation including a respiratory questionnaire, methacholine challenge test with determination of PC20(the provocative concentration that reduced FEV1 by 20% from baseline), exhaled nitric oxide (eNO). Venous blood will be analyzed for complete blood count + eosinophils, IGE levels, hs-CRP. All measurements will be evaluated in a single 3 hour visit, with no follow up study visits.

Primary end point: hs-CRP levels as add on tool to predict negative or positive MCT in children Secondary outcome parameters: All other parameters are the secondary end points.

ELIGIBILITY:
Inclusion Criteria:

* Age range 6 to 18 years
* Patient referred for Methacholine Challenge Test (MCT)

Exclusion Criteria:

* Base line FEV1(forced expiratory volume in the first second) < 65%
* The presence of other systemic or lung disease
* Anti-inflammatory drugs
* Upper respiratory tract infection in the last month

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: subjects (age range 6 to 18 years) referred for Methacholine Challenge Test (MCT)
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
HIgh sensitive C-reactive protein | participants will be followed for the duration of hospital visit, an average of 3 hours
  in peripheral Blood count

SECONDARY OUTCOMES:
Metacholine Challenge Test | participants will be followed for the duration of hospital visit, an average of 3 hours
  As assessed by methacholine challenge test with determination of PC20.
IgE | participants will be followed for the duration of hospital visit, an average of 3 hours
  in peripheral Blood count
complete blood count | participants will be followed for the duration of hospital visit, an average of 3 hours
  in peripheral Blood count
Fractional Exhaled NO | participants will be followed for the duration of hospital visit, an average of 3 hours
  determination of exhaled NO in Exhaled breath
body mass index | participants will be followed for the duration of hospital visit, an average of 3 hours

REFERENCES:
- [Derived] Livnat G, Yoseph RB, Nir V, Hakim F, Yigla M, Bentur L. Evaluation of high-sensitivity serum CRP levels compared to markers of airway inflammation and allergy as predictors of methacholine bronchial hyper-responsiveness in children. Lung. 2015 Feb;193(1):39-45. doi: 10.1007/s00408-014-9658-6. Epub 2014 Oct 21. PMID 25331535